CLINICAL TRIAL: NCT06135818
Title: Same Day Diagnosis of Extrapulmonary TB (TB Serositis and TB Meningitis).
Acronym: Epi-TB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: European Union (Other); Zambart (Other); Biomedical Research and Training Institute (Other); Leiden University Medical Center (Other); University of Cape Town Lung Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Epi-TB
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tuberculosis, Extrapulmonary
Keywords: Tuberculosis; Interferon-gamma; Tuberculosis diagnostics
MeSH Terms: conditions — Tuberculosis, Extrapulmonary; Tuberculosis

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspected extrapulmonary tuberculosis (Experimental): Patients with pleural, pericardial, or peritoneal effusions due to suspected extrapulmonary tuberculosis and those with suspected TB meningitis.
  Interventions: Diagnostic Test: IRISA-TB

INTERVENTIONS:
Diagnostic Test: IRISA-TB — ELISA-based assay that detects interferon-gamma concentrations in extrapulmonary fluid in active TB.

SUMMARY:
Extrapulmonary TB (EPTB) accounts for nearly 30% of TB cases in HIV endemic settings, such as South Africa. The diagnosis of extrapulmonary TB is complicated by the poor performance of Gene Xpert and TB Culture in extrapulmonary fluid (30-50% sensitive), as well as the poor specificity of ADA. We can therefore not reliably use these tests to diagnose EPTB as effectively as we use them in sputum samples. The current best practice for diagnosing pleural TB is to perform a pleural biopsy, which is both invasive and costly. A rapid, easy to use test is needed to allow accurate and fast diagnosis of EPTB. Interferon-gamma is released at high concentrations in extrapulmonary fluid in active EPTB. Antrum Biotech has developed the IRISA-TB assay (validated and SAHPRA licenced) for the diagnosis of EPTB.

The study will assess the real-world performance of IRISA-TB compared to ADA, Gene Xpert, and TB Culture when used to diagnose EPTB. We will evaluate IRISA-TB's performance in the following patient groups:

* Suspected TB pleural effusion (n= 650)
* Suspected TB pericardial effusion (n= 280)
* Suspected TB peritonitis (n= 200)
* Suspected TB meningitis (n = 1040) As part of our evaluation, we will ask clinicians who treat these patients to provide their feedback on IRISA-TB. We will ask them to indicate to what extent the IRISA-TB test helped them to make treatment decisions. Finally, we will conduct an economic assessment to determine the true cost of diagnosing and treating EPTB to the health system and patients, and we will determine how IRISA-TB could potentially result in cost savings.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years and over attending health care facility with symptoms of TB.
2. Serosal or CSF fluid sample provided to NHLS with sufficient volume to perform SOC tests + 1ml.
3. Patients in whom extrapulmonary TB is part of the treating clinicians' differential diagnosis.

Exclusion Criteria:

1. Volunteers who refuse to sign informed consent and/or provide clinical details (Proxy consent will be obtained for participants who are incapacitated, with a follow up consent when they have recovered their capacity to consent)
2. Patients with current significant history of substance or alcohol abuse that may impact study visits.
3. Patients who are unable to communicate by telephone or who do not have a current active traceable contact number.
4. Patients not willing to undergo an HIV test.
5. Patients whose fluid sample volumes are insufficient to perform standard of care testing in addition to IRISA-TB
6. Positive sputum GXP within 2 weeks prior to serosal fluid or CSF sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Test-specific performance outcomes | 24 months
  Comparison of sensitivity, specificity, accuracy, predictive values, likelihood ratios, number needed to treat (NNT) and indeterminate rate for the various diagnostic assays (IRISA-TB, ADA, Gene Xpert, TB Culture)

SECONDARY OUTCOMES:
Empiric treatment rates for extrapulmonary TB | 24 months
  Clinicians will be asked to indicate whether IRISA-TB made an impact on treatment decisions. Empiric treatment rates for extrapulmonary TB are high due to poor performance of current diagnostics.
Cost effectiveness | 24 months.
  Determining the true cost to the health system of various diagnostic strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Aliasgar Esmail, MD FCP, Principal Investigator — UCT Lung Institute, Centre for lung infection and immunity
Locations (4):
- South Africa (2):
  - University of KwaZulu-Natal, Durban, KwaZulu-Natal
  - University of Cape Town Lung Institute, Cape Town, Western Cape
- Zambart, Lusaka, Zambia
- Biomedical Research and Training Institute, Harare, Zimbabwe